CLINICAL TRIAL: NCT01701076
Title: An Open, Multicentric Phase II Trial to Evaluate the Efficacy and Safety of Bendamustine, Lenalidomide (Revlimid®) and Dexamethasone (BRd) as 2nd-line Therapy for Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Bendamustine, Lenalidomide (Revlimid®) and Dexamethasone (BRd) as 2nd-line Therapy for Patients With Relapsed or Refractory Multiple Myeloma
Acronym: BRd
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: Celgene Corporation (Industry); Mundipharma Research GmbH & Co KG (Industry); Mundipharma Medical Company (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, PD Dr. Ulrich Mey, PD Dr.med., Kantonsspital Graubünden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU10.041/BRd; 2010-022253-42 (EudraCT Number)
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Myeloma
Keywords: Relapsed / refractory multiple myeloma; 2nd line treatment
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Lenalidomide; Dexamethasone; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine (Experimental): All patients are treated with bendamustine in combination with lenalidomide and dexamethasone for a maximum of 6 cycles.
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — Induction treatment phase (cycle 1-6):
  * Bendamustine 75 mg/m2 i.v day 1 and 2
  * Lenalidomide 25 mg p.o. day 1-21
  * Dexamethasone 40/20 mg p.o., day 1, 8, 15, 22
  * Pegfilgrastim 6 mg s.c., day 3 in case of severe neutropenia
  Maintenance treatment phase (cycles 7-18):
  * Lenalidomide 25 mg p.o. day 1-21
  * Dexamethasone 40/20 mg p.o., day 1, 8, 15, 22
  Other Names: Lenalidomide; Dexamethasone; Pegfilgrastim

SUMMARY:
Almost all patients with multiple myeloma who survive initial treatment will eventually relapse and require further therapy.

Background: Treatment with lenalidomide and dexamethasone has proven efficacy in two large randomized trials (MM-009 and MM-010) leading to a time to progression (TTP) of 17.1 months for patients with only one prior therapy and a TTP of 10.6 months for 2 and more prior therapies, respectively [1-3]. Continuous treatment with lenalidomide and dexamethasone until disease progression is therefore considered a standard therapy for second line treatment in multiple myeloma patients. However, only a relatively low rate of high quality response (CR, complete response and VGPR, very good partial response) is achieved. High quality responses are associated with with improved progression-free survival and overall survival [4].

Trial: The aim of this trial is to improve high quality response rates for patients with relapsed or refractory multiple myeloma in the 2nd line treatment. This aim shall be achieved by the addition a third anti-myeloma drug (bendamustine) to the established backbone of lenalidomide/ dexamethasone.

Treatment regimen:

* Induction Treatment Phase: Cycles 1-6 Bendamustine 75mg/m2/d day 1 and 2, lenalidomide 25mg/d 1-21, dexamethasone 40mg / 20mg (for patients > 75years) d 1, 8, 15, 22.
* Maintenance Treatment Phase: Cycles 7-18 lenalidomide 25mg/d 1-21, dexamethasone 40mg / 20mg (for patients > 75 years) d 1, 8, 15, 22.

Due to hematoxicity of bendamustine and lenalidomide, administration of pegfilgrastim is mandatory in the induction treatment phase (BRd-regimen)for all patients experiencing severe neutropenia.

The aim of this study is to achieve high quality response rates (CR, VGPR) of ≥ 40%. If this aim is achieved, the treatment of bendamustine in combination with the established lenalidomide/ dexamethasone regimen will be considered promising.

Besides efficacy, the safety of this three-drug regimen is evaluated in this trial.

DETAILED DESCRIPTION:
Assessments for efficacy / response evaluation:

* M-protein quantitation in serum and 24 h urine collection samples by serum- and urine protein electrophoresis
* Quantitation of immunoglobulin levels by nephelometry
* Serum and urine immunofixation
* Free light chain concentrations and ratio in the serum
* Plasma cell percentage in the bone marrow by conventional cytology and biopsy with immunohistochemistry
* Radiologic assessments of the skeleton

Response criteria: Response will be assessed according to IMWG criteria

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients with first relapsed or refractory multiple myeloma (including patients with relapse after high dose chemotherapy followed by autologous stem cell transplantation) who have received no more than one prior line of anti-myeloma treatment
* Treatment with a lenalidomide/ dexamethasone-based 2nd-line regimen is indicated and intended
* Measurable disease as defined by at least one of the following 3 measurements

  * serum monoclonal protein level ≥ 1 g/dl (≥ 10 g/l) or
  * urine M-protein level ≥ 200 mg/24hours or
  * serum FLC assay: Involved FLC level ≥ 10 mg/dl (≥ 100 mg/l) provided serum FLC ratio is abnormal
* ECOG performance status 0, 1, or 2
* Age ≥ 18 years
* All previous cancer therapy (except corticosteroid therapy), including radiation, cytostatic therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
* No prior treatment with a bendamustine-containing regimen allowed
* Prior treatment with lenalidomide is allowed if the treatment is completed > 12 month prior to study entry and the patient responded to prior lenalidomide treatment
* Adequate hematological values:

  * absolute neutrophil count ≥ 1.5 x 109/L
  * platelets ≥ 100 x 109/L
  * hemoglobin > 80 g/L, unless considered to be caused by the underlying hematologic malignancy, based on the investigator's clinical judgement
* Adequate hepatic function:

  * total bilirubin < 1.2 mg/dL
  * AST (SGOT) ≤ 2.5 x ULN
* Adequate renal function:

  o calculated creatinine clearance > 50 ml/min, according to the formula of Cockcroft-Gault
* Disease free of prior malignancies for > 5 years unless the patient

  * has been treated with a curative intent and is considered to be in complete remission for ≥2 years prior to study enrolment
  * or has a curatively-treated

    * basal cell/ squamous cell carcinoma of the skin,
    * carcinoma "in situ"of the cervix,
    * ductal breast carcinoma in situ with complete surgical resection (i.e. negative margins),
    * medullary or papillary thyroid tumor
    * or low grade, early stage localized prostate cancer treated surgically with curative intent

Exclusion Criteria:

* Pregnant or breast feeding females
* Any prior use of bendamustine
* Patients who are unable or unwillingly to undergo antithrombotic therapy
* Any serious underlying medical condition (at the judgment of the investigator) which impairs the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric disorder)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she would participate in the study or any condition significantly confounding the ability to interpret data from the study, based on the local investigator's judgement
* Severe cardiovascular disease, including myocardial infarction within 6 months before study entry, New York Heart Association Class III or IV heart failure, uncontrolled angina or severe uncontrolled ventricular arrhythmias (≥ Lown 3)
* Use of any other experimental drug or therapy/ treatment in a clinical trial within 30 days prior to trial entry
* Known hypersensitivity to study drug(s) or hypersensitivity to any other component of the study drugs
* Any concurrent antineoplastic therapy with chemotherapeutic agents or biologic agents or radiation therapy
* Any major surgical procedure within 30 days prior to study therapy
* Known chronic hepatitis B or C, known HIV infection
* Jaundice or any other severe damage of the liver parenchyma
* Any contraindication for the treatment with bendamustine, lenalidomide, dexamethasone and / or pegfilgrastim in accordance with the appropriate SmPCs
* Any other concomitant drugs contraindicated for use with the study drugs according to the national health authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Efficacy (combined CR-/VGPR-rate) achieved during the induction treatment phase or within four weeks after the last administration of six induction cycles of the BRd regimen | Every 4 weeks up to 7 months

SECONDARY OUTCOMES:
Objective response rates (sCR, CR, VGPR, PR, MR) | Every 4 weeks up to 7 months
Best response (sCR, CR, VGPR, PR, MR) | Every 4 weeks up to 36 months
Time to progression (TTP) | Every 4 weeks up to 36 months
Overall survival (OS) | Every 8 weeks up to 36 months
Safety and tolerability | Every 4 weeks until 30 days after completion of study treatment
  * Type, frequency, severity, and relationship of adverse events to study therapy
  * According to NCI CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mey, MD, Study Chair — Kantonsspital Graubünden
Locations (1):
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Dimopoulos MA, Chen C, Spencer A, Niesvizky R, Attal M, Stadtmauer EA, Petrucci MT, Yu Z, Olesnyckyj M, Zeldis JB, Knight RD, Weber DM. Long-term follow-up on overall survival from the MM-009 and MM-010 phase III trials of lenalidomide plus dexamethasone in patients with relapsed or refractory multiple myeloma. Leukemia. 2009 Nov;23(11):2147-52. doi: 10.1038/leu.2009.147. Epub 2009 Jul 23. PMID 19626046
- [Background] Harousseau JL, Attal M, Avet-Loiseau H. The role of complete response in multiple myeloma. Blood. 2009 Oct 8;114(15):3139-46. doi: 10.1182/blood-2009-03-201053. Epub 2009 Jul 28. PMID 19638622
- [Background] Lentzsch S, O'Sullivan A, Kennedy RC, Abbas M, Dai L, Pregja SL, Burt S, Boyiadzis M, Roodman GD, Mapara MY, Agha M, Waas J, Shuai Y, Normolle D, Zonder JA. Combination of bendamustine, lenalidomide, and dexamethasone (BLD) in patients with relapsed or refractory multiple myeloma is feasible and highly effective: results of phase 1/2 open-label, dose escalation study. Blood. 2012 May 17;119(20):4608-13. doi: 10.1182/blood-2011-12-395715. Epub 2012 Mar 26. PMID 22451423
- [Background] Pönisch W, Heyn S, Wagner I, et al. Combined Bendamustine, Prednisolone and Lenalidomide (RBP) In Refractory or Relapsed Multiple Myeloma. First Results of a Phase I Clinical Trial. Blood, Nov 2010; 116: 1971